CLINICAL TRIAL: NCT03955185
Title: A Non-randomized Controlled Study of Minimally Invasive Versus Abdominal Radical Hysterectomy for Cervical Cancer
Brief Title: Clinical Trial of Minimally Invasive Surgery Versus Abdominal Surgery in Patients With Early Stage Cervical Cancer
Acronym: CGOG 002
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ding Ma, chief physician, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-Surgery1
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-10

CONDITIONS: Uterine Cervical Neoplasm
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive surgery (Experimental): The patients will receive laparoscopic or robotic assisted radical hysterectomy with improved surgery details: 1) Uterine manipulator type Cup-shaped uterine manipulator is prohibited, uterus hanging wire is allowed. 2) Avoid tumor cells shedding into the pelvis: A. Cut the vagina with the transvaginal method, B. Cut the vagina after closed loop ligation of the vagina. After the surgery, they will receive adjuvant therapy according to the pathological risk factors refer to the 2018 NCCN guidelines.
  Interventions: Procedure: minimally invasive surgery
- Open abdominal surgery (Active Comparator): The patients will receive traditional radical hysterectomy.After the surgery, they will receive adjuvant therapy according to the pathological risk factors refer to the 2018 NCCN guidelines.
  Interventions: Procedure: open abdominal surgery

INTERVENTIONS:
Procedure: minimally invasive surgery — Laparoscopic or robotic assisted radical hysterectomy
  Arms: Minimally invasive surgery
Procedure: open abdominal surgery — Traditional open abdominal radical hysterectomy
  Arms: Open abdominal surgery

SUMMARY:
Cervical cancer is the most common cause of death from gynecological cancer world-wide. With technological innovation, minimally invasive or even non-invasive medical treatment has become a trend. Since the first cases of laparoscopic radical hysterectomy of cervical cancer have been reported in 1992, many single-center observational cohort studies have shown that compared to open abdominal surgery ，minimally invasive surgery (laparoscopic or robotic radical hysterectomy) showed advantages of less blood loss, shorter hospital stay and fewer intraoperative complications, while the 5-year survival and disease-free survival were similar. The NCCN guidelines and ESGO recommendations also clearly indicated that patients with FIGO stage IA2 -IIA cervical cancer could undergo open or laparoscopic/robotic radical hysterectomy. However, in October 2018, the results of two studies published in the《New England Journal of Medicine》have subverted our traditional perception of minimally invasive surgery and caused widespread controversy in the field of gynecologic oncology treatment. Both studies showed that the survival rate in the minimally invasive surgery group was lower than that in the open surgery group.

The results of these two studies have brought unprecedented doubts and challenges to the minimally invasive surgery for cervical cancer. The MD Anderson Cancer Center has even stopped minimally invasive surgery for cervical cancer. Several hospitals in Hong Kong have responded similarly. The NCCN guidelines are also quickly updated based on the results of those studies: patients should be informed of the results of this study and doctors should respect the patient's choices. The above research results have also attracted the attention of many gynecological oncologists in the mainland China. Some experts questioned the design of this study design as well as surgical skills. We need to look at these findings cautiously. So, we launched a real-world study of clinical outcomes affected by different surgical treatment for patients of early stage cervical cancer. We plan to recruit 2000 patients with early cervical cancer from 20-30 selected surgical centers nationwide and perform surgery on patients with qualified and experienced doctors.We will inform the patients current status of the study in detail, divide the patients into different observational group according to their choices on surgical methods. The patients will be followed up closely after surgery. We will compare the differences in clinical outcomes between the two surgical methods and conduct subgroup and stratified analysis. We hope that this study can truly reflect the actual status and clinical l level of early cervical cancer treatment in China, and provide a high level of clinical evidence for the treatment of cervical cancer in China .

DETAILED DESCRIPTION:
The study is a non-randomized, prospective, multi-center, clinical study.Patients with early cervical cancer who were enrolled will be divided into two groups: minimally invasive surgery group (group A) and open abdominal surgery group (group B) according to the patient's choice on surgical methods.We will standardize the surgery details according to the factors that may affect the prognosis of cancer treatment in the minimally invasive surgery of cervical cancer, such as : emphasizing the tumor-free principle of surgery; using a ligation band to tighten the vagina before cutting the vagina; avoiding the use of the cup-shaped uterine manipulator；reducing frequent changes in CO2 abdominal pressure；or using a laparoscope-assist transvaginal hysterectomy and other methods to avoid the risk of tumor tissue shedding. Patients with high risk factors after surgery will receive follow-up treatment according to the 2018 NCCN guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FIGO stage (2018) IA1 (with lymph vascular space invasion), IA2, IB1, IB2 or IIA1 disease
* Preoperative histologically confirmed primary adenocarcinoma, squamous cell carcinoma or adenosquamous carcinoma of the uterine cervix
* Age ≤ 65 years old;
* Physical grading: Karnofsky score ≥ 60 points;
* Initial treatment;
* Voluntarily joined the study, signed informed consent, willing to comply, and cooperative with follow-up; (Note: The maximum diameter of the cervical lesion is subject to MRI measurements)

Exclusion Criteria for Preoperative Patients:

* Patients with contraindications to surgery；
* Patients who have previously received pelvic/abdominal radiation or chemotherapy；Patients who had received radiotherapy and chemotherapy for other cancers in the past.
* Patients with evidence of extra cervical metastases by CT, MRI or PET.
* Unable or unwilling to sign informed consent.
* Unable or unwilling to comply with research requirements.
* Patients with diameter of lymph node metastasis ≥ 2 cm by preoperative MRI.
* Patients with pregnancy.
* Patients requiring fertility-preserving surgery.
* Patients who had previously received subtotal hysterectomy.
* Patients participating in other clinical trials.
* Patients with other reasons not suitable clinical trials identified by researchers.

Exclusion Criteria for Postoperative Patients:

* Postoperative pathology: endometrioid adenocarcinoma, clear cell carcinoma, special type adenocarcinoma, neuroendocrine carcinoma (small cell carcinoma), tuberculosis.
* Postoperative tumor size ≥ 4 cm.
* Patients with abdominal aortic lymph node metastasis.
* Patients with severe postoperative complications that are not suitable for adjuvant therapy and affect patient follow-up.
* Patients who did not follow requirements for various reasons (except for various complications and deaths caused by tumor recurrence and metastasis).
* Situation which researchers believe that treatment should be terminated.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) of 3 years | 3 years
  DFS was definite as the time from surgery to disease recurrence
overall survival (OS) of 5 years | up to 5 years
  OS was defined as time from surgery to death by any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, MD;PHD, Study Chair — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
The individual participants data will be preserved in the hospital, and all the chemical or physical examination results will be kept in the medical records, the researches, ethics committee and the drug administration will be permitted to look up all the records as we planned. And all the reports or papers about this research will not relate to the patients' identity. But we do not decide whether the information be available to others, the final decision maybe decided by all the patients in this research.